CLINICAL TRIAL: NCT04309864
Title: Refinement of the Comprehensive Mobile Assessment of Pressure (CMAP) System for Prevention of Pressure Injuries
Brief Title: CMAP Refinement for Pressure Injury Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: B3222-R
Record Dates: First submitted 2020-03-13; First posted 2020-03-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pressure Ulcer
Keywords: skin ulcer; wounds and injuries; decubitus ulcer; wheel chairs; spinal cord injury; seating; pressure injury prevention
MeSH Terms: conditions — Pressure Ulcer; Skin Ulcer; Wounds and Injuries; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Initially, Veteran focus groups will inform researchers regarding needed device refinements; clinician focus groups will inform regarding app updates; then participants will trial the updated seating app for usability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Focus group-Veteran (No Intervention): Veterans will inform study staff regarding desired device design refinements
- Focus group-Clinicians (No Intervention): Clinicians will inform study staff regarding desired app design changes
- Usability-inpatients (Other): Clinicians will use the updated CMAP system during patient education for prevention of pressure injuries with Veterans with SCI who are completing their initial rehabilitation.
  Interventions: Device: Use of CMAP app for education (in-hospital)
- Usability-in-home (Other): The Veteran will use the CMAP system at home for two weeks to use in their daily routines, along with wearing the acti-graph one week prior, two weeks during and one week after CMAP usage.
  Interventions: Device: Use of CMAP app (in-home)

INTERVENTIONS:
Device: Use of CMAP app for education (in-hospital) — Clinicians will use the updated CMAP system during patient education for prevention of pressure injuries with Veterans with SCI who are completing their initial rehabilitation.
  Arms: Usability-inpatients
Device: Use of CMAP app (in-home) — The Veteran will use the CMAP system at home for two weeks during their daily routines.
  Arms: Usability-in-home

SUMMARY:
For Veterans with spinal cord injury who use a wheelchair, pressure injuries related to sitting are a significant daily threat to well-being. Pressure injuries are costly to treat, negatively impact quality of life and community participation, and can be life threatening. Moving or shifting at regular intervals in the wheelchair redistributes harmful pressure and reduces risk for skin breakdown, yet these movements are a challenge to perform consistently. The challenge exists due to lack of sensation to let the individual know they need to shift their weight. Pressure mapping provides a detailed visual representation of pressure distribution and can compensate for impaired sensation. Pressure mapping feedback delivered on-demand on mobile platforms can potentially increase effectiveness in carrying out behaviors to reduce risk for pressure injury when used during clinician-delivered education to set goals and monitor progress and when used at home as a self-management strategy.

DETAILED DESCRIPTION:
Objectives: The long-term goal of this project is to improve the effectiveness of pressure injury prevention education by clinicians and self-management by Veterans with spinal cord injury (SCI) through a methodical development and testing of a mobile platform based pressure mapping system called "Comprehensive Mobile Assessment of Pressure" (CMAP). The targeted risk-reduction behavior in this project is the effective use of weight shifts when sitting in a wheelchair by improving consistency, frequency, duration, and quality of movements to redistribute pressure. CMAP provides visual cues as well as individually customizable reminders that are designed to compensate for the lack of sensation that prevents the use of natural cues to redistribute pressure, by wheelchair users. An updated CMAP system will serve two important objectives: 1) assist clinicians in assessment, individualized goal-setting, and monitoring the Veteran with SCI's progress toward pressure injury prevention behavior goals while in the hospital setting; and 2) assist clinicians with individualized setup and education of the Veteran with SCI for using the CMAP system in the home setting as a self-management strategy for pressure injury prevention.

Specific Aims: The specific aims of this study include: 1a) hardware expansion to improve functionality of the CMAP system to add a docking and charging station and use of CMAP on a smartwatch based on Veteran preferences and 1b) software expansion to enhance clinical education for pressure injury prevention education, with requirements provided by clinicians; 2) determine usability of the refined CMAP system when it is integrated into patient education for Veteran's with acute SCI during their inpatient rehabilitation stay, and 3) a determine usability and efficacy of the refined CMAP system for clinician-delivered pressure injury prevention education, followed by Veteran use of CMAP in their daily routines at home.

Study Design: This four-year study will have multiple stages and will use a mixed methods approach that includes iterative focus groups and interviews with Veterans who have SCI and with clinicians who provide pressure injury prevention education to Veterans with SCI; self-efficacy and usability surveys for both Veterans and clinicians; pilot testing of CMAP during inpatient rehabilitation and testing during outpatient visits. Repeated measures will be used to evaluate changes within subject for completion of weight shifts while using CMAP, compared to periods when not using CMAP.

Methods: During the first two years, improvements to CMAP hardware and software will be guided by experience-based design guided requirements learned about through iterative focus groups including Veterans with SCI/D (n=10) and clinicians (n=10). Usability will be measured at each iteration of development using the System Usability Scale (SUS) and the User Experience Questionnaire (UEQ). The focus groups will be repeated to ensure alignment between development progress and the requirements identified by the focus groups. During the inpatient pilot test, clinician (n=3) and Veteran (n=6) self-efficacy will be measured. Veterans will complete selected sub-scales from the Skin Care Belief Scale and clinicians will answer survey questions developed specifically around providing education for performing weight shifts effectively. Veteran progress toward weight shift goals will be measured through performance monitoring within the CMAP app; Actual performance will be assessed against the individualized goals set by the clinician. During the outpatient testing, Veterans (n=20) will use CMAP at home for 2 weeks after receiving education and individualized goals for weight shift performance by clinicians. While at home, trunk movements will be monitored via actigraphy to monitor weight shift frequency to compare to baseline trunk movement data, weight shift performance data within CMAP app, and finally, compared with individualized goals for performing weight shifts. Self efficacy and usability (SUS and UEQ) of the overall system in both settings will be measured.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1a:

* Veteran adults aged 18-80
* male and female
* with a spinal cord injury (C4 and below) or spinal cord disorder with impaired sensory function and a wheelchair user for at least one year

For Aim 2: Veteran adults aged 18-80, male and female, with a recent spinal cord injury (C4 and below) or a spinal cord disorder with impaired sensory function, who are currently in inpatient rehabilitation with at least 1 week prior to discharge. Participants must demonstrate ability to access the CMAP system application on a mobile phone or tablet independently.

For Aim 3:

* Veteran adults aged 18-80
* male and female
* manual or power wheelchair users
* at least one year post SCI onset
* (C4 and below) or a spinal cord disorder with impaired sensory function
* who are visiting the MVAHCS SCI/D Center for their annual visit or at end of a non-pressure injury stay in the hospital
* at which time review of pressure injury prevention and assessment of wheelchair seating are routinely conducted by clinicians
* Veterans using the CMAP system must demonstrate ability to access the CMAP app on a mobile phone or tablet independently

Clinicians inclusion Criteria for Aim 1b; Aims 2 and 3:

* Clinicians (SCI/D Physical and Occupational Therapists and Nurses and Ancillary Clinician) who, in their normal scope of work, provide patient education for pressure injury prevention

Exclusion Criteria:

For Aim 1a:

* Any Veteran with SCI/D who is unable to verbally and cognitively communicate with the study team

For Aims 2, and 3:

* Any Veteran with SCI/D who has an active pressure injury that contacts their seating system or within six months of a flap surgery
* Any Veteran with SCI/D who is unable to verbally and cognitively communicate with the study team
* Any Veteran whose seat cushion is a customized immersion style

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Usability as measured by System Usability Scale (SUS) | Year 1-2: Change from baseline to second and third focus group
  Aim 1a: The System Usability Scale (SUS) is a 10-item Likert scale (5-item ranging from strongly disagree to strongly agree) which will allow the participants (Veterans) to give their subjective assessment of the Smart watch as part of the CMAP system. Analysis will use Linear Mixed Effects Regression Model
Usability as measured by User Experience Questionaire (UEQ) | Year 1-2: Change from baseline to second and third focus group
  Aim 1a: The User Experience Questionnaire (UEQ) is a 26 -item semantic differential arranged on six scales (attractiveness, perspicuity, efficiency, dependability, stimulation, and, novelty) which will measure the participant's (Veterans) impression of the of their experience with the Smart watch as part of the CMAP system. Analysis will use Linear Mixed Effects Regression Model.
Change in Usability as measured by System Usability Scale (SUS) | Year 1-2: Change from baseline to second and third focus group
  Aim 1b:The System Usability Scale (SUS) is a 10-item Likert scale (5-item ranging from strongly disagree to strongly agree) which will allow the participants (clinicians) to give their subjective assessment of the newly developed educational formats in the CMAP system. Analysis will use Linear Mixed Effects Regression Model
Change in Usability as measured by User Experience Questionaire (UEQ) | Year 1-2: Change from baseline to second and third focus group
  Aim 1b:The User Experience Questionnaire (UEQ) is a 26 -item semantic differential arranged on six scales (attractiveness, perspicuity, efficiency, dependability, stimulation, and, novelty) which will measure the participants' (clinicians) impression of the of their experience with the newly developed educational formats of the CMAP system. Analysis will use Linear Mixed Effects Regression Model.
Change in Usability as measured by System Usability Scale (SUS) | Year 2-3: compare final focus group score to after using in rehabilitation
  Aim 2: The System Usability Scale (SUS) is a 10-item Likert scale (5-item ranging from strongly disagree to strongly agree) which will allow the participants (clinicians) to give their subjective assessment of the educational formats in the CMAP system after using it for Veterans' acute rehabilitation. Analysis will use Linear Mixed Effects Regression Model
Change in Usability as measured by User Experience Questionaire (UEQ) | Year 2-3: compare final focus group score to after using in rehabilitation
  Aim 2: The User Experience Questionnaire (UEQ) is a 26 -item semantic differential arranged on six scales (attractiveness, perspicuity, efficiency, dependability, stimulation, and, novelty) which will measure the participants' (clinicians) impression of the of their experience with the CMAP educational formats after using it for Veterans' acute rehabilitation. Analysis will use Linear Mixed Effects Regression Model.
Change in Usability as measured by System Usability Scale (SUS) | Year 2-3: compare final focus group score to after using in rehabilitation
  Aim 2: The System Usability Scale (SUS) is a 10-item Likert scale (5-item ranging from strongly disagree to strongly agree) which will allow the participants (Veterans) to give their subjective assessment of the CMAP system after using it during their acute rehabilitation. Analysis will use Linear Mixed Effects Regression Model
Change in Usability as measured by User Experience Questionaire (UEQ) | Year 2-3: compare final focus group score to after using in rehabilitation
  Aim 2: The User Experience Questionnaire (UEQ) is a 26 -item semantic differential arranged on six scales (attractiveness, perspicuity, efficiency, dependability, stimulation, and, novelty) which will measure the participants' (Veterans) impression of the of their experience with the CMAP system after using it during Veterans' during their acute rehabilitation. Analysis will use Linear Mixed Effects Regression Model.
Change in Usability as measured by System Usability Scale (SUS) | Year 4: compare initial and final use in the out patient and home setting
  Aim 3: The System Usability Scale (SUS) is a 10-item Likert scale (5-item ranging from strongly disagree to strongly agree) which will allow the participants (clinicians) to give their subjective assessment of the educational formats in the CMAP system after using it for Veterans' in the outpatient and community-based settings . Analysis will use Linear Mixed Effects Regression Model.
Change in Usability as measured by User Experience Questionaire (UEQ) | Year 4: compare initial and final use in the home setting
  Aim 3:The User Experience Questionnaire (UEQ) is a 26 -item semantic differential arranged on six scales (attractiveness, perspicuity, efficiency, dependability, stimulation, and, novelty) which will measure the participants' (clinicians) impression of the of their experience with the CMAP educational formats at the start of intervention and after using the CMAP system in the outpatient and community-based settings. Analysis will use Linear Mixed Effects Regression Model.
Change in Usability as measured by System Usability Scale (SUS) | Year 4: compare initial and final use in the home setting
  Aim 3: The System Usability Scale (SUS) is a 10-item Likert scale (5-item ranging from strongly disagree to strongly agree) which will allow the participants (Veterans) to give their subjective assessment of the CMAP system after using it in the outpatient and community-based settings. Analysis will use Linear Mixed Effects Regression Model.
Change in Usability as measured by User Experience Questionaire (UEQ) | Year 4: compare initial and final use in the home setting
  Aim 3:The User Experience Questionnaire (UEQ) is a 26 -item semantic differential arranged on six scales (attractiveness, perspicuity, efficiency, dependability, stimulation, and, novelty) which will measure the participants' (Veterans) impression of the of their experience with the CMAP system at the start of intervention and after using the CMAP system in the outpatient and community-based settings . Analysis will use Linear Mixed Effects Regression Model.

SECONDARY OUTCOMES:
Change in Self-Efficacy as measured by Skin Care Belief Scale | Year 2-3: Pre post use of the CMAP system
  Aim 2: The Skin Care Belief Scale (King 2012) self efficacy portion (21-items) will be used to measure the participants' (Veterans) perception of pressure injury risk and beliefs about performance of weight shifts. Baseline measure pre-instruction using the CMAP and post-instruction and use of the CMAP system. The responses are scaled: 1= strongly disagree to 5= strongly agree. Analysis will use Linear Mixed Effects Regression Model
Change in Self-Efficacy as measured by customized scale | Year 2-3: Pre post use of the CMAP system
  Aim 2: This self-efficacy measures clinician confidence in delivering pressure injury prevention education, specifically around instruction of how to perform weight shifts using the CMAP system during Veterans' acute rehabilitation. Baseline measure pre-instruction using the CMAP and post-instruction and use of the CMAP system. Analysis will use Linear Mixed Effects Regression Model
Change in Self-Efficacy as measured by Skin Care Belief Scale | Year 4: Pre post use of the CMAP system
  Aim 3: The Skin Care Belief Scale (King 2012) self efficacy portion (21-items) will be used to measure the participants' (Veterans) perception of pressure injury risk and beliefs about performance of weight shifts. Baseline measure pre-instruction using the CMAP and post-use of the CMAP system. The responses are scaled: 1= strongly disagree to 5= strongly agree. Analysis will use Linear Mixed Effects Regression Model
Change in Self-Efficacy as measured by customized scale | Year 4: Pre post use of the CMAP system
  Aim 3: This self-efficacy measures clinician confidence in delivering pressure injury prevention education, specifically around instruction of how to perform weight shifts using the CMAP system during Veterans' acute rehabilitation. Baseline measure pre-instruction using the CMAP and post-use of the CMAP system in the outpatient and home settings. Analysis will use Linear Mixed Effects Regression Model
Weight Shift bout comparisons | Year 4
  Aim 3: Comparing Veteran weight shift activity (measured by actigraphy) pre and post use of CMAP system in the outpatient and community-based settings.

CONTACTS AND LOCATIONS:
Overall Officials: Byron W Eddy, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN; Christine M. Olney, BSN MS PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request, per VA requirements.
Supporting Information: Study Protocol, ICF
Time Frame: At the completion of the study.
Access Criteria: Upon request once the study data analysis are completed and published.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT04309864/ICF_000.pdf